CLINICAL TRIAL: NCT04598126
Title: Effects of Patient Education Manual on Pain, Range of Motion and Function in Patient With Knee Osteoarthritis
Brief Title: Patient Education Manual on Patients With Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCRS/20/1005 Samiah Sarwar
Record Dates: First submitted 2020-10-19; First posted 2020-10-22 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Knee Osteoarthritis
Keywords: Patient education manual; Knee O.A; Pain; ROM
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy (Active Comparator): Traditional physical therapy
  Interventions: Other: Traditional physical therapy
- patient education manual +traditional physical therapy (Experimental): Patient education manual +traditional physical therapy
  Interventions: Other: patient education manual +traditional physical therapy

INTERVENTIONS:
Other: Traditional physical therapy — Traditional physical therapy Ultrasound posteriorly 6 mints 4 days/week hydrocollateral pack anteriorly 10 mints 4 days/week Quadriceps isometrics 10 repetitions×1 set, 4 days/week and Hamstring muscle strechings 10 repetitions×1 set, 4 days/
  Arms: Traditional physical therapy
Other: patient education manual +traditional physical therapy — Patient educational Manual
  + Traditional physical therapy Ultrasound posteriorly 6 mints 4 days/week hydrocollateral pack anteriorly 10 mints 4 days/week Quadriceps isometrics 10 repetitions×1 set, 4 days/week and Hamstring muscle strechings 10 repetitions×1 set, 4 days/
  Arms: patient education manual +traditional physical therapy

SUMMARY:
This RCT was conducted to see effects of patient education manual on pain, ROM and functional performance in patient of knee osteoarthritis. In this study the investigators were provide an educational manual as a home plan in which the investigators educate and guide patients about proper posture, life style modification, precautions and safety measures and home exercise in patient with knee osteoarthritis

DETAILED DESCRIPTION:
This RCT was conducted to see effects of patient education manual on pain, ROM and functional performance in patient of knee osteoarthritis. In this study the investigators provide an educational manual as a home plan in which they educate and guide patients about proper posture, life style modification, precautions and safety measures and home exercise in patient with knee osteoarthritis.

The investigators will divide the patients in two groups. One group was treated with the patient education manual and routine physical therapy and the other group was treated with routine physical therapy alone. After baseline assessment patient was assessed at 2nd, 4th and 6th week and then do final assessment to analyse our results on SPSS, either patient education manual is helpful in minimising there pain functional limitation and increasing their Range Of Motion. Visual analogue scale, goniometry and WOMEC was used to measure outcome regarding pain, Range of motion and functional performance in patients with knee osteoarthritis. This study was help full in the management, to improve function and to decrease status of disability in future in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria

* Idiopathic knee OA-I, II, &III

Exclusion Criteria:

* Post Traumatic OA Knees
* Ligament instability
* Condromalacia patellae
* Knee replacements
* Cognitive impairment
* Rheumatoid arthritis
* Meniscus injury

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale(VAS) | 4th day
  The VAS is a unidimensional measure of pain intensity.it is a continuous scale comprised of a horizontal (HVAS) or vertical (VAS) line, usually 10 centimeters (100 mm) in length. the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 )[100-mm scale]).

SECONDARY OUTCOMES:
WOMAC osteoarthritis index | 4th day
  It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
  * Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
  The WOMAC parameters are:
  0-none,1-slight,2-moderate,3-sever,4-extreme.

OTHER OUTCOMES:
ROM Knee flexion ( Flexion Rt) | 4th day
  Changes from the Baseline ROM range of Motion of knee flexion was taken with the Help of Goniometer
ROM Knee flexion ( Flexion Lt) | 4th day
  Changes from the Baseline ROM range of Motion of knee flexion was taken with the Help of Goniometer
ROM knee Extension ( extension Rt) | 4th day
  Changes from the Baseline ROM range of Motion of knee extension was taken with the Help of Goniometer
ROM knee extension ( extension Lt) | 4th day
  Changes from the Baseline ROM range of Motion of knee extension was taken with the Help of Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur-Rehman, Principal Investigator — Riphah International University
Locations (1):
- Rehabilitation department CMH(Combined military hospital), Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iqbal MN, Haidri FR, Motiani B, Mannan A. Frequency of factors associated with knee osteoarthritis. J Pak Med Assoc. 2011 Aug;61(8):786-9. PMID 22356003
- [Background] Lespasio MJ, Piuzzi NS, Husni ME, Muschler GF, Guarino A, Mont MA. Knee Osteoarthritis: A Primer. Perm J. 2017;21:16-183. doi: 10.7812/TPP/16-183. PMID 29035179
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Loeser RF. Aging and osteoarthritis: the role of chondrocyte senescence and aging changes in the cartilage matrix. Osteoarthritis Cartilage. 2009 Aug;17(8):971-9. doi: 10.1016/j.joca.2009.03.002. Epub 2009 Mar 12. PMID 19303469
- [Background] Liaqat M, Liaqar B, Rauf R, Bashir F. Prevalence of knee osteoarthritis and quality of life in middle aged adults. International Journal of Rehabilitation Sciences (IJRS). 2018;7(02):26-8.
- [Background] Wallace IJ, Worthington S, Felson DT, Jurmain RD, Wren KT, Maijanen H, Woods RJ, Lieberman DE. Knee osteoarthritis has doubled in prevalence since the mid-20th century. Proc Natl Acad Sci U S A. 2017 Aug 29;114(35):9332-9336. doi: 10.1073/pnas.1703856114. Epub 2017 Aug 14. PMID 28808025
- [Background] Plotnikoff R, Karunamuni N, Lytvyak E, Penfold C, Schopflocher D, Imayama I, Johnson ST, Raine K. Osteoarthritis prevalence and modifiable factors: a population study. BMC Public Health. 2015 Nov 30;15:1195. doi: 10.1186/s12889-015-2529-0. PMID 26619838
- [Background] Pal CP, Singh P, Chaturvedi S, Pruthi KK, Vij A. Epidemiology of knee osteoarthritis in India and related factors. Indian J Orthop. 2016 Sep;50(5):518-522. doi: 10.4103/0019-5413.189608. PMID 27746495
- [Background] Sowers M, Karvonen-Gutierrez CA, Jacobson JA, Jiang Y, Yosef M. Associations of anatomical measures from MRI with radiographically defined knee osteoarthritis score, pain, and physical functioning. J Bone Joint Surg Am. 2011 Feb 2;93(3):241-51. doi: 10.2106/JBJS.I.00667. PMID 21266638
- [Background] Jarvholm B, Lewold S, Malchau H, Vingard E. Age, bodyweight, smoking habits and the risk of severe osteoarthritis in the hip and knee in men. Eur J Epidemiol. 2005;20(6):537-42. doi: 10.1007/s10654-005-4263-x. PMID 16121763
- [Background] Stubbs B, Aluko Y, Myint PK, Smith TO. Prevalence of depressive symptoms and anxiety in osteoarthritis: a systematic review and meta-analysis. Age Ageing. 2016 Mar;45(2):228-35. doi: 10.1093/ageing/afw001. Epub 2016 Jan 20. PMID 26795974
- [Background] Rashan L, Hamidpour R. OsteoLuban a Novel Natural Remedy for Osteoarthritis. 2019.
- [Background] Creamer P, Lethbridge-Cejku M, Hochberg MC. Where does it hurt? Pain localization in osteoarthritis of the knee. Osteoarthritis Cartilage. 1998 Sep;6(5):318-23. doi: 10.1053/joca.1998.0130. PMID 10197166
- [Background] Farrokhi S, Chen YF, Piva SR, Fitzgerald GK, Jeong JH, Kwoh CK. The Influence of Knee Pain Location on Symptoms, Functional Status, and Knee-related Quality of Life in Older Adults With Chronic Knee Pain: Data From the Osteoarthritis Initiative. Clin J Pain. 2016 Jun;32(6):463-70. doi: 10.1097/AJP.0000000000000291. PMID 26308705
- [Background] Sharma L. Local factors in osteoarthritis. Curr Opin Rheumatol. 2001 Sep;13(5):441-6. doi: 10.1097/00002281-200109000-00017. PMID 11604602
- [Background] van Tunen JAC, Peat G, Bricca A, Larsen LB, Sondergaard J, Thilsing T, Roos EM, Thorlund JB. Association of osteoarthritis risk factors with knee and hip pain in a population-based sample of 29-59 year olds in Denmark: a cross-sectional analysis. BMC Musculoskelet Disord. 2018 Aug 21;19(1):300. doi: 10.1186/s12891-018-2183-7. PMID 30126395
- [Background] Mora JC, Przkora R, Cruz-Almeida Y. Knee osteoarthritis: pathophysiology and current treatment modalities. J Pain Res. 2018 Oct 5;11:2189-2196. doi: 10.2147/JPR.S154002. eCollection 2018. PMID 30323653